CLINICAL TRIAL: NCT01816672
Title: A Multi-Center, Prospective, Clinical Trial Comparing the Efficacy of AutoloGel Therapy to Usual and Customary Care in Wagner 1 and 2 Diabetic Foot Ulcers
Brief Title: Efficacy of AutoloGel Therapy to Usual and Customary Care in Wagner gd 1 and 2 Diabetic Foot Ulcers.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Cytomedix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CM001
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Wagner 1; Wagner 2; Non healing diabetic foot wound
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AutoloGel (Active Comparator): AutoloGel treatment
  Interventions: Device: AutoloGel
- Usual and Customary Care (Other): Standard of care
  Interventions: Other: Usual and Customary Care

INTERVENTIONS:
Device: AutoloGel — Treatment with Autologel and standard of care twice a week for the first two weeks and once a week thereafter
  Other Names: Autologel System
  Arms: AutoloGel
Other: Usual and Customary Care — Standard of care treatment twice weekly for 2 weeks then weekly
  Other Names: Standard of care clinically indicated
  Arms: Usual and Customary Care

SUMMARY:
The purpose of this study is to determine if AutoloGel platelet rich plasma used on non healing diabetic foot ulcers Wagner gd. 1 and 2 is more effective then the usual and customary care

DETAILED DESCRIPTION:
Autologel is a platelet-rich plasma gel used in the treatment of no-healing chronic wounds. Prospective observational studies of the effectiveness of Autologel have demonstrated promising results in regard to the healing of diabetic foot ulcers including severe Wagner grade 3 and 4 ulcers. The aim of the current trial is to compare the efficacy, measured as wound healing in a single-blind (assessor) randomized controlled trial, of usual and customary care with and without Autologel in treating Wagner 1 and 2 diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Medicare eligible
2. ≥18 years of age
3. Type I or II diabetes requiring medical treatment as determined by the physician
4. The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (index ulcer) is a Wagner 1 or 2 Diabetic Foot Ulcer (DFU; see Appendix 9 for Wagner Classification) that is located on the plantar, medial, or lateral aspect of the foot (including all toe surfaces but not on the heel). Subjects who have heel ulcers may be included if another, eligible wound is the index ulcer
5. For subjects with potentially multiple eligible DFUs, the largest ulcer will be selected. There must be at least 4 cm between the index ulcer and other ulcers; if all ulcers are closer than 4 cm, the subject should not be enrolled (screen failure)
6. Debrided ulcer size between 0.5 cm2 and 20 cm2
7. Demonstrated adequate offloading regimen
8. Duration ≥ 1 month at first visit (screening period)
9. Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician.

Exclusion Criteria:

1. Subjects known to be sensitive to AutoloGel components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Wagner 3, 4, or 5 DFU (see Appendix 9 for Wagner Classification) Page 15 of 58
3. Any clinically infected index ulcer that is apparent on Day 0. The presence of infection is defined by ≥ 2 classic findings of inflammation (erythema, warmth, tenderness, pain, or induration) or purulent secretions (Lipsky, 2012, or see Appendix 4)
4. Presence of another wound that is concurrently treated and might interfere with index wound
5. Ulcer not of DFU pathophysiology (e.g., venous, vasculitic, radiation, rheumatoid, collagen vascular disease, pressure, or arterial etiology)
6. Presence of underlying osteomyelitis, or if osteomyelitis is suspected
7. Received systemic corticosteroids or immunosuppressive agents, hyperbaric oxygen therapy (HBOT), electrostimulation, growth factors, or any cell or tissue-derived products for wounds during the 30 days preceding the screening visit; received radiation therapy or chemotherapy within previous 6 months
8. Any malignancy other than non-melanoma skin cancer
9. Ischemic ulcer defined as an ankle brachial index (ABI; handheld or Arterial Doppler) < 0.8 (note: if ABI is ≥ 1, then an skin perfusion pressure (SPP) or transcutaneous oximetry (TCOM) must be performed or the subject cannot be enrolled), TCOM < 30 mm Hg, or SPP < 30 mm Hg; toe pressure < 45 mm Hg. These measurements may be concurrent with the initial evaluation of the index ulcer or obtained within 90 days of study enrollment if done prior to that concurrence.
10. Subject has radiographic evidence consistent with diagnosis of active Charcot foot
11. Untreated Charcot foot or DFUs associated with a treated Charcot deformity in which reconstruction or offloading has not taken place
12. Ulcer expected to be treated with any advanced therapeutics (e.g., HBOT)
13. Ulcer area decreases by ≥ 30% during 2-week screening/run-in period
14. Subjects who are cognitively impaired and do not have a healthcare proxy
15. Serum albumin of less than 2.5 g/dL
16. Plasma Platelet count of less than 100 x 109/L
17. Hemoglobin of less than 10.5 g/dL
18. Subject has inadequate venous access for repeated blood draw required for AutoloGel Administration
19. Subject requires or is anticipated to require interventions directed at improvement of arterial perfusion to affected area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Compare time to heal in Wagner 1 and 2 diabetic foot ulcers at 12 weeks treated with AutoloGel versus usual and customary care | 12 weeks
  Complete wound closure is defined as skin re-epithelialization without drainage or dressing requirements confirmed at consecutive study visits 2 weeks apart. Initial diagnosis of healing by unblinding Principal Investigator will be confirmed by an independent blinded observer using digital photography, planimetry data and wound measurements

SECONDARY OUTCOMES:
Assess wound healing trajectory and change in Chronic Wound quality of Life W-QOL scores: and to assess the comparative safety of AutoloGel and usual and customary care | 13 weeks
  QOL tool administered prior to and at the end of treatment to document the impact of the wound on the subject's life and whether treatment interventions helped a return to improved functioning.
Number of patients with adverse events as a measure of tolerability | 12 weeks
  Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Forest General Hospital, Hattiesburg, Mississippi, United States